CLINICAL TRIAL: NCT03499028
Title: Improvement of Patient Satisfaction and Clinical Outcomes Using JointCOACH to Manage the Episode of Care for THA and TKA Bundles
Brief Title: Improvement of Patient Satisfaction and Clinical Outcomes Using JointCOACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-063
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (No Intervention): The Standard of Care Group will receive standard, routine medical care and will communicate with their surgeon and clinical care team through conventional methods such as phone.
- Experimental (JointCOACH) Group (Experimental): The Experimental Group will receive standard, routine medical care and utilize a web-based communication platform called JointCOACH to communicate with their care team via computer or smartphone throughout their episode of care. They will also receive information personalized to their treatment plan and will be asked to complete online questionnaires.
  Interventions: Other: JointCOACH

INTERVENTIONS:
Other: JointCOACH — Patients randomized to this group will utilize JointCOACH to communicate with their surgical team, receive information
  Arms: Experimental (JointCOACH) Group

SUMMARY:
JointCOACH is a web-based communication platform that enables joint replacement patients to communicate with their care team via computer or smartphone throughout their episode of care, from the time that surgery is scheduled until at least 90 days postoperatively.

DETAILED DESCRIPTION:
Patients will receive the following information at key intervals: 1) instructions about how to prepare for surgery, 2) information about the procedure, 3) information about medications and pain control, 4) information about postoperative recovery and rehabilitation. In addition, several surveys will be distributed using JointCOACH to keep patients involved in their own recovery and to keep the surgical team informed of their progress. The proposed research will help determine if JointCOACH can improve patient satisfaction and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary total hip or primary total knee arthroplasty
* Willing to sign an IRB approved informed consent form
* Have internet access or mobile access with a valid email address at the time of enrollment
* Above the age of 18 years

Exclusion Criteria:

* Staged arthroplasty procedure within 6 months of the index procedure
* Abandoned email address of record (e.g. bounce of email from clinic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Higuera, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Visperas AT, Greene KA, Krebs VE, Klika AK, Piuzzi NS, Higuera-Rueda CA. A Web-Based Interactive Patient-Provider Software Platform Does Not Increase Patient Satisfaction or Decrease Hospital Resource Utilization in Total Knee and Hip Arthroplasty Patients in a Single Large Hospital System. J Arthroplasty. 2021 Jul;36(7):2290-2296.e1. doi: 10.1016/j.arth.2021.01.037. Epub 2021 Jan 21. PMID 33581971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period - May 2018 - March 2020 Recruitment location - single large academic healthcare system
Pre-assignment Details: Patients were consented and randomized into the standard of care (SOC) or JointCOACH group during the same visit. Since patients were randomized at time of consent, those that eventually had cancelled surgeries were removed from the Total Started in Participant Flow.
Period: Overall Study
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Started | 226 | 220
Completed | 204 | 195
Not Completed | 22 | 25
Not completed — Lost to Follow-up | 12 | 9
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Unplanned SNF discharge | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group | Total
Number analyzed (Participants) | 204 | 195 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 66 (9) | 65 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 102 | 215
  Male | 91 | 93 | 184
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 195 | 189 | 384
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 204 | 195 | 399
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.04 (5.9) | 31.48 (2.85) | 31.76 (5.83)
Age-Adjusted Charlson Comorbidity Index [Mean (Standard Deviation); unit: index score] — Age-adjusted Charlson Comorbidity Score is derived by the summation of the weighted scores of 19 medical conditions found to be associated with survival and age. The lower the score the healthier the patient. The higher the score, the higher morbidity. Range is from 0-37.
  index score | 2.67 (1.6) | 2.85 (1.7) | 2.75 (1.62)
Education Level [Count of Participants; unit: Participants]
  Did Not Complete High School | 2 | 0 | 2
  High School | 47 | 47 | 94
  Some College | 58 | 64 | 122
  Bachelor's Degree | 57 | 43 | 100
  Master's Degree | 26 | 26 | 52
  Advanced | 14 | 15 | 29
Employment Status [Count of Participants; unit: Participants]
  Unemployed | 11 | 6 | 17
  Employed | 84 | 76 | 160
  Homemaker | 1 | 5 | 6
  Retired | 108 | 108 | 216
ASA Classification [Count of Participants; unit: Participants] — The American Society of Anesthesiologists Physical Status Classification (ASA I to ASA VI) grades patients on their perioperative risk. Examples of ASA classifications include: ASA I - a normal healthy patient, ASA III - a patient with severe systemic disease, ASA V- a moribund patient who is not expected to survive without the operation.
  Participants
    I | 1 | 2 | 3
    II | 67 | 68 | 135
    III | 133 | 123 | 256
    IV | 3 | 2 | 5
Diagnosis [Count of Participants; unit: Participants]
  Osteoarthritis | 190 | 188 | 378
  Osteonecrosis | 9 | 3 | 12
  Post-traumatic Osteoarthritis | 3 | 1 | 4
  Rheumatoid Arthritis | 0 | 1 | 1
  Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Picker Patient Experience (PPE-15) Questionnaire
Description: It is a 15-item patient experience questionnaire. Each response will be categorized as a problem or non-problem and reported as the percent of respondents reporting a problem, averaged across all PPE-15 domains.
Time Frame: 30 and 90 days after index surgery
Measure: Mean (Standard Deviation); unit: percentage of problem responses
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Number analyzed (Participants) | 204 | 195
percentage of problem responses
  30 days after index surgery | 13 (18) | 13 (18)
  90 days after index surgery | 11.1 (16) | 12.3 (17)

2. Secondary Outcome: Visual Analog Scale (VAS) for Patient Satisfaction
Description: It is a satisfaction measurement tool using a scale from 0-100, where 0 = completely dissatisfied and 100 = completely satisfied.
Time Frame: 30 and 90 days after index surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Number analyzed (Participants) | 204 | 195
score on a scale
  30 days after index surgery | 94.2 (12.4) | 93.6 (10.6)
  90 days after index surgery | 94.2 (11.1) | 94.7 (9.9)

3. Secondary Outcome: Length of Hospital Stay
Description: It is a count of the number of days the patient was admitted to the hospital after the index procedure prior to being discharged (measured in days)
Time Frame: 90 days after index surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Number analyzed (Participants) | 204 | 195
days | 1.4 (0.8) | 1.5 (0.8)

4. Secondary Outcome: Discharge Disposition
Description: Number of patient routinely discharged to home
Time Frame: 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Number analyzed (Participants) | 204 | 195
Participants | 199 | 187

5. Secondary Outcome: Number of Participants With Readmissions
Description: It is a count of the number patients with hospital readmissions related to the index procedure within 30 and 90 days after the index procedure.
Time Frame: 30 and 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Number analyzed (Participants) | 204 | 195
Participants
  30 days after surgery | 0 | 1
  90 days after surgery | 2 | 3

6. Secondary Outcome: Number of Participants With Reoperations
Description: It is a count of the number of reoperations related to the index procedure within 30 and 90 days after the index procedure.
Time Frame: 30 and 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Number analyzed (Participants) | 204 | 195
Participants
  30 days after surgery | 0 | 0
  90 days after surgery | 0 | 0

7. Secondary Outcome: Number of Subjects With Emergency Department Visits
Description: It is a count of the number of subjects with emergency department visits related to the index procedure within 30 and 90 days after the index procedure.
Time Frame: 30 and 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Number analyzed (Participants) | 204 | 195
Participants
  30 days after surgery | 0 | 1
  90 days after surgery | 0 | 1

8. Secondary Outcome: Number of Outpatient Follow-Up Visits
Description: It is a count of the number of outpatient follow-up visits with the surgical team related to the index procedure within 30 and 90 days after the index procedure.
Time Frame: 30 and 90 days after index surgery
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Number analyzed (Participants) | 204 | 195
visits
  30 days after surgery | 0.80 (0.49) | 0.80 (0.55)
  90 days after surgery | 1.79 (0.56) | 1.84 (0.6)

9. Secondary Outcome: Number of Telephone Calls
Description: It is a count of the number of telephone calls with the surgical team related to the index procedure within 30 and 90 days after the index procedure.
Time Frame: 30 and 90 days after index surgery
Measure: Mean (Standard Deviation); unit: calls
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
Number analyzed (Participants) | 204 | 195
calls
  30 days after surgery | 1.28 (1.61) | 1.31 (1.58)
  90 days after surgery | 2.03 (2.15) | 2.06 (2.25)

10. Secondary Outcome: Provider Satisfaction Survey- JointCOACH Satisfaction
Description: It is a 2 question survey regarding provider experience using JointCOACH measured using a 5-point Likert scale, where 1 = very dissatisfied and 5 = very satisfied.
Time Frame: 90 days after the last patient enrolled has had surgery. approximately 22 months after the first patient enrolled. All study-related intervention is complete at this time.
Population: Providers - Surgeon (n=4), Physician Assistant (n=2), Nurse Practitioner (n=1), Nurse (n=3). Providers were not considered enrolled but did contribute to this assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Provider Satisfaction: For this outcome, providers were asked about their satisfaction with JointCOACH. No arms were designated for this outcome.
Arm/Group | Provider Satisfaction
Number analyzed (Participants) | 10
Participants
  Very Unsatisfied | 0
  Unsatisfied | 0
  Neutral | 3
  Satisfied | 5
  Very Satisfied | 2

11. Secondary Outcome: Provider Satisfaction Survey- JointCOACH Recommendation
Description: as for outcome 10
Time Frame: 90 days after the last patient enrolled has had surgery. All study-related intervention is complete at this time.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Groups:
- Provider Satisfaction: For this outcome, providers were asked about whether they would recommend the use of JointCOACH. No arms were designated for this outcome.
Arm/Group | Provider Satisfaction
Number analyzed (Participants) | 10
Participants
  Very Unlikely | 0
  Unlikely | 0
  Neutral | 4
  Likely | 4
  Very Likely | 2

ADVERSE EVENTS:
Time Frame: 3 month period after surgery
Description: Adverse events were manually collected
Arm/Group | Standard of Care Group | Experimental (JointCOACH) Group
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/195
Serious Adverse Events (participants affected / at risk) | 2/204 | 1/195
Other Adverse Events (participants affected / at risk) | 0/204 | 0/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Group (N=204) | Experimental (JointCOACH) Group (N=195)
Manipulation Under Anesthesia (Musculoskeletal and connective tissue disorders) | 2 | 1 — Manipulation Under Anesthesia is done to increase range of motion after total joint arthroplasty.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03499028/Prot_SAP_000.pdf